CLINICAL TRIAL: NCT04173520
Title: ELRIAH Score: A Simple Score for HCC Risk Stratification in CHC Patients With Cirrhosis or Advanced Liver Fibrosis Who Achieved SVR Following DAA Therapy
Status: Completed | Type: Observational
Sponsor: Egyptian Liver Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SCORE
Record Dates: First submitted 2019-11-17; First posted 2019-11-22 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: HCC
MeSH Terms: interventions — bis(p-chlorophenyl)acetic acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: DDA — Follow up after SVR

SUMMARY:
aimed to develop a scoring system to assess risk of developing HCC in a large cohort of chronic hepatitis C (CHC) patients with advanced hepatic fibrosis (F3) or cirrhosis (F4) with sustained virological response (SVR) after receiving direct acting antivirals (DAAs).

DETAILED DESCRIPTION:
Current guidelines recommend biannual surveillance for hepatocellular carcinoma (HCC) in all patients with cirrhosis. However, risk of HCC incidence is not the same for different patients. The study aimed to develop a scoring system to assess risk of developing HCC in a large cohort of chronic hepatitis C (CHC) patients with advanced hepatic fibrosis (F3) or cirrhosis (F4) with sustained virological response (SVR) after receiving direct acting antivirals (DAAs).

ELIGIBILITY:
Inclusion Criteria:

* no history of previous HCC
* SVR after DAAs treatment

Exclusion Criteria:

* history of previous HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2326 CHC patients (638 patients with F3 and 1734 with F4 stage)
Sampling Method: Non-Probability Sample
Enrollment: 2326 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Rate of HCC incidence after viral clearance | 12-45 months after SVR

IPD SHARING:
Plan to Share IPD: No